CLINICAL TRIAL: NCT07404553
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II/III Study to Evaluate the Efficacy and Safety of SHR-1918 in Patients With Hypercholesterolemia With Inadequate Lipid Control on Statins Plus PCSK9 Inhibitors
Brief Title: A Study Of SHR-1918 In Participants With Hypercholesterolemia With Inadequate Lipid Control on Statins Plus PCSK9 Inhibitors
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1918-303
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1918 Injection Group (Experimental): SHR-1918 injection.
  Interventions: Drug: SHR-1918 Injection
- SHR-1918 Injection Placebo Group (Placebo Comparator): SHR-1918 injection placebo.
  Interventions: Drug: SHR-1918 Injection Placebo

INTERVENTIONS:
Drug: SHR-1918 Injection — SHR-1918 injection.
  Arms: SHR-1918 Injection Group
Drug: SHR-1918 Injection Placebo — SHR-1918 injection placebo.
  Arms: SHR-1918 Injection Placebo Group

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of SHR-1918 in patients with hypercholesterolemia with inadequate lipid control on statins plus PCSK9 inhibitors. The efficacy and safety of SHR-1918 will be evaluated after 12-weeks and 24-weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ≥ 18 years old and ≤ 85 years old, who is able and willing to provide a written informed consent.
2. TG ≤ 5.6 mmol/L.
3. LDL-C ≥ 2.6 mmol/L for moderate to high ASCVD risk, LDL-C ≥ 1.8 mmol/L for very high ASCVD risk, LDL-C ≥ 1.4 mmol/L for ultra-high ASCVD risk.
4. Male and female subjects of childbearing potential and their partners must have no plans to donate sperm or become pregnant during the entire study period and after the last dose, and agree to use contraceptive methods as specified in the protocol.

Exclusion Criteria:

1. History of severe allergies/hypersensitivity reactions, or clinically significant allergies/hypersensitivity reactions as judged by the investigator, or history of allergies to drugs with similar chemical structures.
2. Heart failure with New York Heart Association (NYHA) Class III-IV prior to screening or randomization.
3. Acute ischemic ASCVD events within 3 months prior to screening or randomization.
4. Have severe cardiac arrhythmia within 3 months prior to screening or randomization.
5. Echocardiography indicates a left ventricular ejection fraction (LVEF) of less than 30% within 3 months prior to screening.
6. History of percutaneous coronary intervention, history of coronary artery bypass grafting (CABG), history of peripheral arterial revascularisation within 1 month prior to screening or randomization.
7. Poorly controlled type 2 diabetes mellitus or previously diagnosed type 1 diabetes mellitus; poorly controlled hypertension.
8. Have a history of diseases that significantly affect blood lipid levels, such as nephrotic syndrome, severe liver diseases, Cushing's syndrome, or have severe arrhythmia prior to screening or randomization.
9. Malignant tumors within 5 years.
10. It's planned to research transcutaneous coronary intervention, coronary artery bypass grafting, carotid or peripheral artery reconstruction, pacemaker implantation, cardiac resynchronisation therapy (CRT), implantable cardioverter defibrillator (ICD) implantation and other implantations during the study.
11. Received plasma exchange therapy within 2 months prior to screening, or plans to receive plasma exchange therapy during the study period, or has received LDL receptor gene therapy prior to screening.
12. Have a history of major surgery within 3 months prior to screening, or plans to undergo major surgery during the study period.
13. History of drug use, substance abuse, and alcohol abuse.
14. Participated in or is participating in other clinical studies and has received study interventions within the past month prior to screening.
15. Researchers determine that the subject has poor compliance or any factors that make them unsuitable for participation in this trial, including but not limited to participation in the study placing the subject at unacceptable risk or potentially interfering with the study results.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Percentage change in low density lipoprotein cholesterol (LDL-C) levels at Week 12 relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Percentage change in low density lipoprotein cholesterol (LDL-C) levels at Week 24 relative to baseline. | At 24 weeks of treatment.
  Phase 3.

SECONDARY OUTCOMES:
Percentage change in non-high-density lipoprotein cholesterol (non-HDL-C) relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Percentage change in triglyceride (TG) relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Percentage change in total cholesterol (TC) relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Percentage change in apolipoprotein B (ApoB) relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Percentage change in Apolipoprotein A1 (ApoA1) relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Change in triglyceride (TG) relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Change in non-high-density lipoprotein cholesterol (non-HDL-C) relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Change in total cholesterol (TC) relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Change in apolipoprotein B (ApoB) relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Change in Apolipoprotein A1 (ApoA1) relative to baseline. | AT 12 weeks of treatment.
  Phase 2.
Change in Lipoprotein(a) (Lp(a)) relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Percentage change in Lipoprotein(a) (Lp(a)) relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Change in high-density lipoprotein cholesterol (HDL-C) relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Percentage change in high-density lipoprotein cholesterol (HDL-C) relative to baseline. | At 12 weeks of treatment.
  Phase 2.
Proportion of subjects with the overall LDL-C achievement rate. | At 12 weeks of treatment.
  Phase 2.
Proportion of subjects with the LDL-C achievement rates in different risk groups. | At 12 weeks of treatment.
  Phase 2.
Change in LDL-C decreased by ≥ 50% to baseline. | At 12 weeks of treatment.
  Phase 2.
Percentage change in LDL-C decreased by ≥ 50% to baseline. | At 12 weeks of treatment.
  Phase 2.
Incidence and severity of adverse events (AEs). | Approximately 12 weeks.
  Phase 2.
Incidence and severity of injection site reactions. | Approximately 12 weeks.
  Phase 2.
Percentage change in non-HDL-C relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Percentage change in TG relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Percentage change in TC relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Percentage change in ApoB relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Percentage change in ApoA1 relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Change in TG relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Change in non-HDL-C relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Change in TC relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Change in ApoB relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Change in ApoA1 relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Change in Lp(a) relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Percentage change in Lp(a) relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Change in HDL-C relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Percentage change in HDL-C relative to baseline. | At 24 weeks of treatment.
  Phase 3.
Proportion of subjects with the overall LDL-C achievement rate. | At 24 weeks of treatment.
  Phase 3.
Proportion of subjects with the LDL-C achievement rates in different risk groups. | At 24 weeks of treatment.
  Phase 3.
Change in LDL-C decreased by ≥ 50% to baseline. | At 24 weeks of treatment.
  Phase 3.
Percentage change in LDL-C decreased by ≥ 50% to baseline. | At 24 weeks of treatment.
  Phase 3.
Incidence and severity of adverse events (AEs). | Approximately 24 weeks.
  Phase 3.
Incidence and severity of injection site reactions. | Approximately 24 weeks.
  Phase 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided